CLINICAL TRIAL: NCT06530004
Title: Clinical Follow-up Study of Rituximab in the Treatment of Nephrotic Syndrome in Children
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bai Haitao, MD, Director, The First Affiliated Hospital of Xiamen University
Other Study IDs: XDFY-EK-BHT
Record Dates: First submitted 2024-06-14; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Nephrotic Syndrome; Rituximab; Children; Efficacy
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Rituximab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sequential prevention group: According to the situation of B cells to rebuild the preventive use of rituxan, each 375 mg/m2.
  Interventions: Drug: Rituximab
- Recurrent sequential group: In patients with recurrence after the use of rituxan, each 375 mg/m2.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — B lymphocyte reconstitution was performed regularly after the administration of rituximab, and 1-4 doses of rituximab were given according to the exhaustion of B cells in children.

SUMMARY:
This was a retrospective study. Children who were diagnosed with refractory nephrotic syndrome and treated with rituximab (RTX) and followed up for ≥1 year in the Department of Pediatrics, the First Affiliated Hospital of Xiamen University from March 2020 to March 2026 were enrolled. Personal information, past medical history, clinical examination data and follow-up data before and after the use of RTX were extracted from the medical record system. (1) The median relapse-free survival, the number of relapses and the adverse reactions of RTX were compared before and after RTX treatment, and the clinical efficacy and safety of RTX were evaluated. (2) By comparing the annual relapse frequency, reduction and withdrawal of steroids and immunosuppressive agents, B cell reconstitution and adverse drug reactions between prophylactic RTX and post-relapse RTX maintenance regimens; (3) Multivariate analysis of risk factors for recurrence of nephropathy after RTX treatment. (4) growth indicators monitoring patient evaluation and RTX medical economic benefit analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children clinically diagnosed with FRNS/SDNS/SRNS with complete clinical data;
* age < 18 years old;
* For the first time using RTX treatment, and used in nephrotic syndrome ease;
* The follow-up for 1 year or more.

Exclusion Criteria:

* Congenital or infantile nephrotic syndrome, secondary nephrotic syndrome (such as lupus nephritis, IgA nephropathy, purpura nephritis, hepatitis B nephritis, etc.);
* Active stage of hepatitis, complicated with severe infection, severe deficiency of immune response, malignant diseases;
* Estimated glomerular filtration rate (GFR) <60mL/min/1.73m2.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who were diagnosed with refractory nephrotic syndrome and treated with rituximab (RTX) and followed up for ≥1 year in the Department of Pediatrics, the First Affiliated Hospital of Xiamen University from March 2020 to March 2026 were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The median relapse-free survival | 1 year
  The median relapse-free survival of nephrotic syndrome before and after RTX treatment was compared.
Different sequential group curative effect evaluation | 1 year
  After comparing the preventive RTX and recurrence RTX maintain annual recurrent treatment。

SECONDARY OUTCOMES:
Risk factors for renal disease recurrence after RTX treatment. | 1 year
  Multivariate cox analysis was used to analyze the risk factors of relapse after rituximab treatment in children with nephrotic syndrome by including gender, age of onset of nephrotic syndrome, course of disease before rituximab, history of immunosuppressive therapy, age of rituximab treatment, and maintenance immunosuppressive therapy after rituximab.

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of xiamen university, Xiamen, Fujian, China